CLINICAL TRIAL: NCT06840080
Title: Short-term Effect of Oleoylethanolamide (OEA) and LipiSperse Supplementation on Metabolic Pathways in Otherwise Healthy Participants - a Single Blind, Cross-over Study
Brief Title: OEA and LipiSperse Metabolic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Gencor Pacific Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: GLP1PK
Record Dates: First submitted 2025-01-22; First posted 2025-02-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers - Male and Female; Pharmacokinetic Study in Healthy Volunteers
Keywords: Healthy volunteer; OEA; oleoylethanolamide
MeSH Terms: interventions — oleoyl ethanolamine; oleoylethanolamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Single dose of 2 capsules will be administered that appear identical to active arms.
  Interventions: Other: Placebo
- 125mg OEA with LipiSperse (Experimental): Single dose of 2 capsules will be administered. 1 capsule will contain 125mg OEA and 13.9mg of LipiSperse and 1 capsule will be a placebo.
  Interventions: Dietary Supplement: 125mg OEA with LipiSperse
- 250mg OEA with LipiSperse (Experimental): Single dose of 2 capsules will be administered. Each capsule will contain 125mg OEA and 13.9mg of LipiSperse.
  Interventions: Dietary Supplement: 250mg OEA with LipiSperse

INTERVENTIONS:
Other: Placebo — Single dose of 2 capsules. Capsules contain the same excipients as the active arms, except for the OEA with LipiSperse in capsules that appear identical to the OEA with LipiSperse capsules
  Arms: Placebo
Dietary Supplement: 125mg OEA with LipiSperse — Single dose of 2 capsules. 1 capsule contains 125mg of OEA and 13.9mg of LipiSperse, the other capsule is a placebo.
  Other Names: 125mg oleoylethanolamide
  Arms: 125mg OEA with LipiSperse
Dietary Supplement: 250mg OEA with LipiSperse — Single dose of 2 capsules. Each capsule contains 125mg of OEA and 13.9mg of LipiSperse.
  Other Names: 250mg oleoylethanolamide
  Arms: 250mg OEA with LipiSperse

SUMMARY:
A placebo controlled, single blind, cross-over study evaluating the short-term effect of oleoylethanolamide (OEA) with LipiSperse supplementation on metabolic pathways in healthy participants.

DETAILED DESCRIPTION:
This study aims to compare the metabolic effects of two different doses of OEA with LipiSperse to a placebo in healthy participants over an 8-hour period. There are three trial arms in this study. Each participant will complete all 3 arms of the study, for a 3-way cross-over.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 years and older
* Generally healthy
* BMI 25.0-34.9 kg/m2
* Able to provide informed consent
* Agree to not participate in another clinical trial while enrolled in this trial
* Agree not to change current diet and/or exercise frequency or intensity during entire study period
* Females using a prescribed form of birth control (e.g. oral contraceptive)
* Participant's ability to participate fully and comply with demands of the study including attendance at all scheduled blood collection time points

Exclusion Criteria:

* Have a serious illness e.g. neurological disorders such as MS, kidney disease, liver disease or heart conditions
* History of any glucose or insulin regulation problem, including diabetes.
* Have an unstable illness e.g. thyroid gland dysfunction, uncontrolled mood disorders (e.g., depression, anxiety, bipolar).
* Diagnosed with any known metabolic or endocrine dysfunctions e.g., diabetes, NAFLD, hyperinsulinemia, hypoglycaemia.
* Use of any medication or supplements that may affect any metabolic pathway associated with satiety (e.g., GLP-1, GIP, glucagon), glucose or insulin.
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Significant change in diet in the past 1-month (e.g., removal of a food group or calorie restriction)
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>21 alcoholic drinks week)
* Pregnant or lactating women
* Allergic to any of the ingredients in active or placebo formula
* Participants who are or who have participated in any other clinical trial during the past 1 month (excludes RDC clinical trials which are to be assessed on a case-by-case basis).
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Regular use within the past 4 weeks of supplements containing OEA and/or LipiSperse

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males and Females who are cisgender
Enrollment: 40 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Changes in serum/plasma GLP-1 AUC | Baseline and 8 hours
  Change from baseline to the end of the study period in serum/plasma GLP-1 AUC for each arm of treatment.

SECONDARY OUTCOMES:
Changes in serum/plasma GIP AUC | Baseline and 8 hours
  Change from baseline to the end of the study period in serum/plasma GIP AUC for each of the 3 arms.
Changes in serum/plasma DPP-4 AUC | Baseline and 8 hours
  Change from baseline to the end of the study period in serum/plasma DPP-4 AUC for each of the 3 arms.
Changes in serum/plasma glucagon AUC | Baseline and 8 hours
  Change from baseline to the end of the study period in serum/plasma glucagon AUC for each of the 3 arms.
Changes in serum/plasma glucose AUC | Baseline and 8 hours
  Change from baseline to the end of the study period in serum/plasma glucose AUC for each of the 3 arms.
Changes in serum/plasma insulin AUC | Baseline and 8 hours
  Change from baseline to the end of the study period in serum/plasma insulin AUC for each of the 3 arms.
Tmax of GLP-1 | Baseline to 8 hours
  Tmax of GLP-1 for each of the 3 arms.
Tmax of GIP | Baseline to 8 hours
  Tmax of GIP for each of the 3 arms.
Tmax of DPP-4 | Baseline to 8 hours
  Tmax of DPP-4 for each of the 3 arms.
Tmax of glucagon | Baseline to 8 hours
  Tmax of glucagon for each of the 3 arms.
Tmax of glucose | Baseline to 8 hours
  Tmax of glucose for each of the 3 arms.
Tmax of insulin | Baseline to 8 hours
  Tmax of insulin for each of the 3 arms.
Cmax of GLP-1 | Baseline to 8 hours
  Cmax of GLP-1 for each of the 3 arms.
Cmax of GIP | Baseline to 8 hours
  Cmax of GIP for each of the 3 arms.
Cmax of DPP-4 | Baseline to 8 hours
  Cmax of DPP-4 for each of the 3 arms.
Cmax of glucagon | Baseline to 8 hours
  Cmax of glucagon for each of the 3 arms.
Cmax of glucose | Baseline to 8 hours
  Cmax of glucose for each of the 3 arms.
Cmax of insulin | Baseline to 8 hours
  Cmax of insulin for each of the 3 arms.
Individual absorption data for each subject | Baseline to 8 hours
  Individual change data obtained for serum/plasma GLP-1, GIP, DPP-4, glucagon, glucose and insulin from each participant for each of the 3 study arms will be individually compared for change. Individual results will then be combined for whole group comparison/analysis.
Tolerability including GIT tolerance | Baseline to 8 hours
  Tolerability including Gastrointestinal (GIT) tolerance. A GIT tolerance questionnaire will be administered prior to lunch. Will be reviewed for each of the 3 arms
Safety via AE monitoring | Baseline to 8hours post dose
  Safety via AE monitoring for each of the 3 arms
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (AUC change in GLP-1) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for total AUC change in GLP-1 over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (AUC change in GIP) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for total AUC change in GIP over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (AUC change in DPP-4) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for total AUC change in DPP-4 over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (AUC change in glucagon) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for total AUC change in glucagon over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (AUC change in glucose) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for total AUC change in glucose over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (AUC change in insulin) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for total AUC change in insulin over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (Tmax of GLP-1) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Tmax of GLP-1 over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (Tmax of GIP) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Tmax of GIP over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (Tmax of DPP-4) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Tmax of DPP-4 over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (Tmax of glucagon) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Tmax of glucagon over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (Tmax of glucose) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Tmax of glucose over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (Tmax of insulin) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Tmax of insulin over 8-hours
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (CMax of GLP-1) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Cmax of GLP-1 over 8-hours.
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (CMax of GIP) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for GIP over 8-hours.
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (CMax of DPP-4) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Cmax of DPP-4 over 8-hours.
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (CMax of glucagon) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Cmax of glucagon over 8-hours.
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (CMax of glucose) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Cmax of glucose over 8-hours.
Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used (CMax of insulin) | Baseline to 8 hours
  Non-inferiority/equivalence comparison of the two different OEA and LipiSperse doses used for Cmax of insulin over 8-hours.
VAS for appetite | Baseline to 4 hours
  A visual analogue scale (VAS) for appetite will be administered 3.5 - 4 hours after dosing, and will be assessed for each of the 3 arms.
Food consumption during the time in clinic (Lunch) | Baseline to 8 hours.
  Participants will be supplied with a standardised lunch meal of known nutritional value (i.e., calories, carbohydrate, fat and protein content). Each participants food will be provided to them via a standardised container (i.e., the same dimension with foods segregated). Prior to and upon completion of the meal, all meal containers will be photographed. The photos will be used to assess the percentage of food that was consumed at each of the 3 visits.
Food consumption during the time in clinic (Breakfast) | Baseline to 8 hours.
  Participants will be supplied with a standardised breakfast meal of known nutritional value (i.e., calories, carbohydrate, fat and protein content). Each participants food will be provided to them via a standardised container (i.e., the same dimension with foods segregated). Prior to and upon completion of the meal, all meal containers will be photographed. The photos will be used to assess the percentage of food that was consumed at each of the 3 visits.
Food consumption during the time in clinic (snacks) | Baseline to 8 hours.
  Any snacks consumed during the day (baseline to 8-hours) at each visit will be recorded. The number of snacks consumed during each visit will be assessed as a numerical number (i.e., number of biscuits or pieces of fruit). The difference in snacks consumed at each visit will then be analysed for any differences

OTHER OUTCOMES:
E/LFT for triglycerides, cholesterol and safety markers | Baseline and 8 hours
  Electrolyte/Liver Function Test (E/LFT) for triglycerides, cholesterol and safety markers for each arm. Samples will be analysed for a range of safety biomarkers within the E/LFT including Sodium, Potassium, Chloride, Bicarbonate, Calcium.

CONTACTS AND LOCATIONS:
Overall Officials: Ramasamy Venkatesh, Study Director — Gencor Pacific
Locations (1):
- RDC Clinical, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No